CLINICAL TRIAL: NCT04376450
Title: A Comparative Evaluation of Nonincised Papillae and Entire Papilla Preservation Surgical Approach in the Treatment of Intrabony Defects - a Clinical and Radiographic Study
Brief Title: Nonincised Papillae in the Treatment of Intrabony Defects.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: SVS Institute of Dental Sciences (Other)
Responsible Party: Principal Investigator, Dr R Viswa Chandra, Principal Investigator, SVS Institute of Dental Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SVSIDS/PERIO/2/2018
Record Dates: First submitted 2020-04-29; First posted 2020-05-06 (Actual); Last update posted 2020-05-06 (Actual); Status verified 2020-05

CONDITIONS: Reconstructive Surgical Procedure
Keywords: Periodontitis; reconstructive surgical procedure;; guided tissue regeneration;; surgical flaps;treatment outcome
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Intervention Model Description: GROUP A: NONINCISED PAPILLAE SURGICAL APPROACH (NIPSA) GROUP B: ENTIRE PAPILLA PRESERVATION TECHNIQUE (EPP)
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: a randomized, triple-blinded, parallel study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nonincised Papillae Surgical Approach (Experimental): Nonincised papillae surgical approach is a papillae preservation technique, where an apical approach is carried out, without incisions or disinsertion of tissues at the level of the papillae or marginal tissues.
  Interventions: Procedure: Experimental- Nonincised papillae surgical approach
- Entire Papilla Preservation Technique (Active Comparator): Entire Papilla preservation technique is a tunnel-like procedure to preserve the defect associated papilla
  Interventions: Procedure: Active comparator- Entire papilla preservation technique

INTERVENTIONS:
Procedure: Experimental- Nonincised papillae surgical approach — The basic principle of the technique is the placement of only one buccal horizontal or oblique incision in the mucosa, as apically as possible from the periodontal defect and the marginal tissues, and the raising of a mucoperiosteal flap coronally, which permits apical access to the defect but leaving the marginal tissues intact, acting as a "dome" for the protection of the clot.
  Other Names: NIPSA
  Arms: Nonincised Papillae Surgical Approach
Procedure: Active comparator- Entire papilla preservation technique — The entire Papilla Preservation Technique is to preserve the whole integrity of the defect- associated papilla providing a tunnel-like undermining incision. The completely preserved interdental papilla provides an intact gingival chamber to stabilize the blood clot and improve the wound healing process. To provide adequate access for debridement, EPP requires a short buccal vertical releasing incision on the buccal side of the neighboring tooth extending just beyond the mucogingival line.
  Other Names: EPP
  Arms: Entire Papilla Preservation Technique

SUMMARY:
The primary objective of the present study is to clinically and radiographically evaluate nonincised papillae surgical approach and entire papilla preservation approach for the treatment of intrabony defects with GTR membrane and hydroxyapatite graft.

DETAILED DESCRIPTION:
Various procedures to treat intrabony defects by preserving the interdental papilla include conventional, simplified, and modified papilla preservation techniques. The drawback of these techniques is the post-surgical gingival recession.

In order to overcome this drawback, the "entire papilla preservation" technique has been proposed, by preserving the whole integrity of the defect associated papilla providing a tunnel-like undermining incision. Recently a novel surgical procedure, termed nonincised papillae surgical approach (NIPSA), was designed to maintain the integrity of the interdental soft tissues covering intrabony defects. This would prevent biomaterial exposure associated with loss of papillary height, increase the amount of space for hard and soft tissue regeneration, and minimize gingival recession.

ELIGIBILITY:
Inclusion Criteria:

1. Systemically healthy individuals within an age group 30-60yrs with chronic periodontal disease.
2. Presence of two or more intrabony defects with probing pocket depth ≥5mm, CAL≥5mm, and radiographic depth ≥4mm.
3. Adequate attached gingiva of 3mm and vestibular depth of 8mm. -

Exclusion Criteria:

1. Uncontrolled systemic disease.
2. Pregnancy and lactation.
3. Defects involving lingual sites.
4. Presence of restoration in the experimental teeth.
5. Smokers -

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Estimated)
Dates: Start 2019-03-06 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
CLINICAL ATTACHMENT LEVEL (CAL) | Baseline to 6 months
  measured from the cemento-enamel junction (CEJ) to the bottom of the pocket
POCKET PROBING DEPTH (PPD) | Baseline to 6 months
  from the gingival margin to the bottom of the pocket;
Intrabony component (INTRA) of the defect | Baseline to 6 months
  the distance from the most coronal extension of the interdental bone crest (BC) to the bottom of the defect (BD) (BC-BD).

SECONDARY OUTCOMES:
Papilla loss (PL) | Baseline to 6 months
  measured from contact point to tip of the papilla.
Local bleeding score | Baseline to 6 months
  recorded as positive when bleeding on probing was present at the surgical site.

CONTACTS AND LOCATIONS:
Locations (1):
- R V Chandra, Hyderabad, Telangana, India

IPD SHARING:
Plan to Share IPD: No